CLINICAL TRIAL: NCT05669170
Title: Evaluating Safety and Potential Benefit of Methylphenidate as a Symptomatic Treatment for Apathy in Veterans With Parkinson's Disease.
Brief Title: Methylphenidate for Apathy in Veterans With Parkinson's Disease
Acronym: MAV-PD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Olga Brawman-mintzer, Staff Physician, Ralph H. Johnson VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX002673-01
Record Dates: First submitted 2022-12-16; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease; Apathy
Keywords: methylphenidate; apathy; Parkinson disease
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — Psychosocial Intervention; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Methylphenidate 20 mg
  Interventions: Behavioral: Psychosocial intervention; Drug: Methylphenidate
- Placebo (Placebo Comparator): Placebo
  Interventions: Behavioral: Psychosocial intervention

INTERVENTIONS:
Behavioral: Psychosocial intervention — The counseling session, in which a trained study clinician will counsel the primary caregiver, will take place at each study visit and after the randomization visit. It will last approximately 20-30 minutes. Each counseling session will consist of the following elements:
  * Review and adjustment of the patient and caregiver supportive care plans
  * Emotional support and the opportunity to ventilate feelings
  * Counseling regarding specific caregiving skills
  * Assistance with problem-solving of specific issues that the caregiver brings to the sessions
  * Answers to questions regarding the educational materials The educational materials will consist of a copy of the book "The 36-Hour Day" by Nancy L. Mace and Peter V. Rabins. The caregiver also will be provided with 24-hour phone access to the study nurse or physician for assistance with crises that may arise after hours.
Drug: Methylphenidate — norepinephrine and dopamine reuptake inhibitor
  Arms: Treatment

SUMMARY:
Apathy is one of the most common behavioral symptoms of Parkinson's disease. Patients with apathy show diminution in motivation and goal-directed behaviors, which is a fundamental aspect of human functioning, affecting dependency and quality of life. Although apathy is thought to be potentially treatable currently there are no effective treatments for apathy. Given the higher incidence of medical and psychiatric comorbidities, the Veterans Affairs health system represents a unique population for which medication response may be different from the general population. This study aims to evaluate if a medication that has already been proven to be useful in Alzheimer's disease patients with apathy, could be helpful in Parkinson's disease as well as decreasing its debilitating consequences and reducing patients' dependency on caregivers, providing well-deserved relief to patients and their loved ones.

DETAILED DESCRIPTION:
Apathy in Parkinson's disease (PD) is a significant public health problem with serious adverse consequences for patients and caregivers. Apathy is present in up to 70% of people with PD. Patients suffering from apathy experience decreased motivation, relying heavily on caregivers to initiate daily activities. The presence of apathy is associated with worse quality of life for patients and caregivers. Moreover, patients with apathy have a faster disease progression and increased likelihood of development of cognitive impairment.

Despite the high prevalence of apathy in PD and its serious consequences, there are no proven treatments for this condition. Dopaminergic enhancement appears as a potential mechanism as there is evidence that degeneration of the frontostriatal circuits involving the prefrontal cortex is one of the main mechanisms for the presence of apathy in PD as well as other neurodegenerative disorders, such as Alzheimer's disease (AD). This degeneration is associated with deficits in dopaminergic and noradrenergic input fibers to the prefrontal cortex.

Methylphenidate, a dopamine and noradrenaline reuptake inhibitor, has been shown to be safe and effective in PD in the treatment of motor and cognitive symptoms, and several small trials and case series reported improvement in motivation and mood. Recently, methylphenidate was shown to be safe and improve apathy in AD in a series of well-controlled studies conducted by members of our team. This represents a relevant result as similar pathophysiology for apathy has been suggested in both AD and PD.

Given the common biological pathways in the onset of apathy in both disorders, we propose that, as is the case in AD, methylphenidate will be a safe and effective treatment for apathy in PD.

The goal of the proposed study of Methylphenidate for Apathy in Veterans with Parkinson's Disease (MAV-PD) is to expand upon this encouraging preliminary work by evaluating methylphenidate for the treatment of apathy in PD Veteran patients. It is our strong belief that a trial designed specifically in Veteran population should be conducted, as reliance on data from civilian populations who differ in their level of medical and psychiatric comorbidity, which influence drug response, may not be applicable to Veterans with PD.

This study will employ a single-site, parallel, randomized, double-blind, placebo-controlled design conducted on 60 Veterans with apathy and PD. MAV-PD is designed specifically for PD patients with apathy, and as such it employs a concise battery of neuropsychological tests that have been chosen for this patient group.

This project is of great importance because it will explore the efficacy and safety of a promising dopamine agonist for treating apathy in PD, where there are no proven treatment options. Should methylphenidate be found effective, it will likely become the first-line therapy for apathy in PD.

ELIGIBILITY:
Inclusion Criteria:

* • Clinically established or probable Parkinson disease according to the Movement Disorders Society Clinical Diagnostic Criteria for Parkinson's Disease

  * Age 40 or older at the time of screening
  * Montreal Cognitive Assessment (MoCA) score between 17-30.
  * Clinical Dementia Rating scale (CDR) lower than 1 and CDR sum of boxes lower than 4.5. The CDR is a numeric scale used to quantify the severity of symptoms of dementia. Using a structured interview protocol, qualified raters assess the subject's cognitive and functional performance in six areas: memory, orientation, judgement, and problem solving, community affairs, home and hobbies, and personal care. Scores are combined to obtain a composite score ranging from 0 through 3. A score between 0 and 1 indicates none or mild symptoms. The individual scores can also be added up, which gives the sum of boxes score.
  * Clinically significant apathy for at least four weeks for which either the frequency of apathy as assessed by the Neuropsychiatric Inventory (NPI) is 'Very frequently', or the frequency of apathy as assessed by the NPI is 'Frequently' or 'Often' AND the severity of apathy as assessed by the NPI is 'Moderate' or 'Marked'
  * Provision of informed consent for participation in the study by the patient. The ability to provide consent will be determined by the Assessment of Capacity for Everyday Decision-Making (ACED). The total score must be 9 (out of 10) or higher to meet the criteria for the study.
  * Availability of primary caregiver, who spends greater than ten hours a week with the patient and supervises his/her care, to accompany the patient to study visits and to participate in the study
  * Sufficient fluency of both the patient and caregiver in written and spoken English
  * No change to PD medications within the month preceding randomization, including starting, stopping, or dosage modifications
  * Treatment with stable doses of levodopa and cholinesterase inhibitors (ChEIs) is allowable if stable for 3 months before randomization. Other psychotropics (with the exclusion of antipsychotics), if stable for 3 months, may be allowed only with PIs' approval on a case-by-case basis

Exclusion Criteria:

* • Meets criteria Major Depressive Episode according to the Diagnostic Statistical Manual of Mental Disorder 5

  * History of psychotic symptoms due to another illness (i.e., schizophrenia, psychosis in mood disorders, etc.) in the past 2 years
  * Clinically significant agitation/aggression for which either the frequency of agitation/aggression as assessed by the NPI is 'Very frequently', or the frequency of agitation/aggression as assessed by the NPI is 'Frequently' AND the severity of the agitation as assessed by the NPI is 'Moderate', or 'Marked'
  * Clinically significant delusions for which either the frequency of delusions as assessed by the NPI is 'Very frequently', or the frequency of delusions as assessed by the NPI is 'Frequently' AND the severity of the delusions as assessed by the NPI is 'Moderate', or 'Marked'
  * Clinically significant hallucinations for which either the frequency of hallucinations as assessed by the NPI is 'Very frequently', or the frequency of hallucinations as assessed by the NPI is 'Frequently' AND the severity of the hallucinations as assessed by the NPI is 'Moderate', or 'Marked'
  * Clinically significant impulse control disorders as assessed by the QUIP
  * Substance use disorder in the past year as assessed by the Drug Abuse Screening Test (DAST-10).
  * Treatment with psychotropic medications in the 2 weeks prior to randomization with the exception of approved treatments for cognitive impairment (ChEIs and memantine), selective serotonin reuptake inhibitor antidepressants, and trazodone (if used as an aid to facilitate sleep and not as an antidepressant); other psychotropics (with the exclusion of antipsychotics), if stable for 3 months, may be allowed only with PI approval on a case-by-case basis. Note that antipsychotics are expressly prohibited
  * Treatment with methylphenidate is contraindicated in the opinion of the PIs
  * Failure of treatment with methylphenidate in the past for apathy
  * Treatment with a medication that would prohibit the safe concurrent use of methylphenidate such as monoamine oxidase inhibitors and tricyclic antidepressants
  * Need for acute psychiatric hospitalization
  * Active suicidal ideation as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS).60 If any of the responses to the questionnaires are yes, the subject will be evaluated by a psychiatrist to assess the risk of suicidality.
  * Uncontrolled hypertension (medication non-compliance or past 3 months with a diastolic reading of 105 mmHg)
  * Symptomatic coronary artery disease deemed to be significant by the PIs at the time of screening
  * Unintentional weight loss as determined by the PIs in the last three months
  * Significant communicative impairments that prohibit meaningful participation in the study assessments
  * Current participation in a clinical trial
  * Hyperthyroidism, advanced arteriosclerosis, symptomatic cardiovascular disease, serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, or a family history of sudden death or death related to heart problems
  * Glaucoma, pheochromocytoma, or known or suspected hypersensitivity to methylphenidate or its excipients
  * CNS abnormalities (e.g., cerebral aneurysm) and/or other vascular abnormalities such as vasculitis or pre-existing stroke, motor tics or family history or diagnosis of Tourette's syndrome, seizures (convulsions, epilepsy), or abnormal EEGs
  * Any condition that, in the opinion of the PIs, makes it medically inappropriate or risky for the patient to enroll in the trial
  * Women who are currently pregnant (methylphenidate is category D). Screening will include pregnancy test

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Apathy Evaluation Scale (AES) | 6 weeks
  This measure is an 18-item scale initially developed as a method for measuring apathy resulting from brain-related pathology.
Clinical Global Impression of Change (CGIC) | 6 weeks
  The CGIC is a systematic method, developed for the Alzheimer's disease (AD) setting to assess clinically significant change in a clinical trial as viewed by an independent, skilled, and experienced clinician and has been used as an outcome in Parkinson disease trials

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | 6 weeks
  This scale was developed specifically to assess cognitive functioning in patients with Alzheimer's disease but has also been used in Parkinson disease.65 It is widely used in clinical trials, and its sensitivity in detecting cognitive changes has been demonstrated in a number of studies. Scores are obtained for orientation, word-list recall, and recognition, object naming, ability to follow simple requests, ideational and constructional praxis, and expressive language. Higher scores indicate worse performance.
Continuous Performance Test (CPT) | 6 weeks
  The CPT was developed to study vigilance or selective attention. In its original form, letters were presented to participants visually one at a time at a fixed rate. The subjects were to press a lever whenever the target letter X appeared and to not press the lever if any other letter was shown. This is called the X-CPT version, and Beck et al found that this version had adequate classification accuracy. Various modifications of the basic X-CPT have been adopted, including changing the target to a number or picture, or a letter series. The CPT version used for this study will be Conner's CPT Version II. The targets are letters and patients do not respond to the letter X (not-X-CPT).
Trail Making Test (TMT) | 6 weeks
  The TMT is composed of visual search and sequencing tasks that are heavily influenced by executive functioning (concentration, resistance to distraction, and cognitive flexibility/set-shifting) and attention. These easily administered tasks are extremely sensitive to neuropsychological deficits such as frontal lobe deficits, problems with psychomotor speed, visual search, and sequencing deficits. The Test has two parts: A and B. In Part A, subjects connect numbers in order on a piece of paper as quickly as possible. Part A provides a baseline for processing speed for interpretation of the second part, Part B. For Part B, subjects connect numbers and letters alternately in order such that the connections are 1-A-2-B-3-C and so on. Both parts are timed. Lower times are better.
Neuropsychiatric Inventory (NPI) | 6 weeks
  The NPI assesses the type and severity of behavioral disturbances in dementia. The inventory evaluates 12 domains of neuropsychiatric symptoms (NPS): apathy, agitation, delusions, hallucinations, depression, euphoria, aberrant motor behavior, irritability, disinhibition, anxiety, sleeping, and eating. Frequency (1 = occasionally, less than once/week; 2 = often, about once per week; 3 = frequently, more than once a week; 4 = very frequently, once or more/day or continuously) and severity (1 = mild, 2 = moderate, 3 = severe) scales in each domain are scored based on responses from an informed caregiver involved in the patient's life. The NPI also includes a 5-point rating used to quantify caregiver distress with the patient's NPS symptoms. To obtain an NPI score for each domain, the severity score and the frequency score are multiplied, and the caregiver distress ratings of each domain are added up.
Starkstein Apathy Scale (SAS) | 6 weeks
  The AS consists of 14 items phrased as questions that are to be answered on a four-point Likert scale. Total score range is 0-42; higher scores indicate more severe apathy.This scale is derived from AES and is tailored to PD. It has been widely validated for the use of Apathy in PD and is recommended by the Movement Disorders Society
Dementia Apathy Interview Rating (DAIR) | 6 weeks
  The DAIR is a structured interview administered to a caregiver. The rationale to include in the trial is to maintain consistency with the ADMET trial, which will help with comparison between groups. It consists of 29 questions concerning the initiation of behavior, interest, and engagement with the environment. Each interview question consists of two parts. The first part addresses issues of frequency on a four-point scale, with 0 signaling the absence of the behavior and 3 signaling the constant presence of the behavior. The second part of the question asks if the current behavior represents a change from the behavior prior to memory loss. The apathy score is a sum of all items reflecting change, divided by the number of items completed, with higher scores representing greater average apathy. Dividing by the number of items adjusts for the number of behaviors for which there has been a change and expresses the patient's apathy score in terms of the underlying 4-point scale (0-3).
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 6 weeks
  This measure is an ADL inventory developed by the ADCS to assess functional performance in patients with AD but has also been used in PD. In a structured interview format that requires less than 15 minutes to administer, informants are queried as to whether subjects attempted each of 24 items in the inventory during the prior 4 weeks and their level of performance. The scale discriminates well the stages of severity of patients, from very mild to severely impaired. It has good test-retest reliability. It includes items from traditional basic ADL scales (e.g., grooming, dressing, walking, bathing, feeding, toileting) as well as instrumental activities of daily living scales (e.g., shopping, preparing meals, using household appliances, keeping an appointment, reading). The ADCS-ADL inventory has been used as an outcome measure in other PD clinical trials.
Questionnaire for Impulsive-Compulsive Disorders in PD (QUIP) | 6 weeks
  Impulse control disorders (ICDs) are often seen in association with apathy in PD. Dopaminergic medications are considered one of the main mechanisms for the development of impulse control disorders, such as gambling. Given the NPI does not address ICDs another screening tool needs to be added. The QUIP is a widely used questionnaire used for screening of ICDs, The total QUIP-RS score for all ICDs and related disorders combined ranges from 0 to 112 with higher number indicating more severe and/or frequent impulse control disorders.
Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - Part III and IV | 6 weeks
  The MDS-UPDRS is one of the most commonly used scales to monitor symptoms related to Parkinson disease. Part III focuses on the primary motor aspects of the condition and part IV focuses on motor fluctuations. Higher scores represent more severe symptoms of parkinsonism. The score range from 0 to 108.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mintzer J, Lanctot KL, Scherer RW, Rosenberg PB, Herrmann N, van Dyck CH, Padala PR, Brawman-Mintzer O, Porsteinsson AP, Lerner AJ, Craft S, Levey AI, Burke W, Perin J, Shade D; ADMET 2 Research Group. Effect of Methylphenidate on Apathy in Patients With Alzheimer Disease: The ADMET 2 Randomized Clinical Trial. JAMA Neurol. 2021 Nov 1;78(11):1324-1332. doi: 10.1001/jamaneurol.2021.3356. PMID 34570180
- [Background] Rosenberg PB, Lanctot KL, Drye LT, Herrmann N, Scherer RW, Bachman DL, Mintzer JE, ADMET Investigators. Safety and efficacy of methylphenidate for apathy in Alzheimer's disease: a randomized, placebo-controlled trial. J Clin Psychiatry. 2013 Aug;74(8):810-6. doi: 10.4088/JCP.12m08099. PMID 24021498
- [Background] Le Heron C, Holroyd CB, Salamone J, Husain M. Brain mechanisms underlying apathy. J Neurol Neurosurg Psychiatry. 2019 Mar;90(3):302-312. doi: 10.1136/jnnp-2018-318265. Epub 2018 Oct 26. PMID 30366958
- [Background] Aarsland D, Larsen JP, Lim NG, Janvin C, Karlsen K, Tandberg E, Cummings JL. Range of neuropsychiatric disturbances in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 1999 Oct;67(4):492-6. doi: 10.1136/jnnp.67.4.492. PMID 10486397
- [Background] Pagonabarraga J, Kulisevsky J, Strafella AP, Krack P. Apathy in Parkinson's disease: clinical features, neural substrates, diagnosis, and treatment. Lancet Neurol. 2015 May;14(5):518-31. doi: 10.1016/S1474-4422(15)00019-8. Epub 2015 Apr 12. PMID 25895932